CLINICAL TRIAL: NCT01998035
Title: Phase I/IIa Study of the Oral 5-Azacitidine in Combination With the Histone Deacetylase Inhibitor Romidepsin for the Treatment of Patients With Relapsed and Refractory Lymphoid Malignancies
Brief Title: Romidepsin Plus Oral 5-Azacitidine in Relapsed/Refractory Lymphoid Malignancies
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: PI left institution
Sponsor: Columbia University (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AAAM3752
Record Dates: First submitted 2013-11-20; First posted 2013-11-28 (Estimated); Results first posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Lymphoid Malignancies; Lymphoma; Hodgkin Lymphoma; Non-hodgkin Lymphoma
Keywords: Lymphoid Malignancies; Lymphoma; Hodgkin Lymphoma; Non-hodgkin Lymphoma; Follicular Lymphoma; Diffuse Large B-Cell Lymphoma; Anaplastic Large Cell Lymphoma; Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; Mantle Cell Lymphoma; Marginal Zone Lymphoma; Burkitt Lymphoma; Waldenstrom Macroglobulinemia; Peripheral T-cell Lymphoma; Cutaneous T-cell Lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Lymphoma, Non-Hodgkin; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Anaplastic; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Waldenstrom Macroglobulinemia; Lymphoma, T-Cell, Peripheral; Lymphoma, T-Cell, Cutaneous | interventions — romidepsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- R/O: Level -1 (Experimental): Oral 5-Azacitidine 100 mg (Days 1-14) Romidepsin (10 mg/m2, Day 8), cycle length (28 days)
  Interventions: Drug: RomiDEPsin 10 MG/M2; Drug: Oral 5-Azacitidine 100 MG
- R/O: Level 1 (Experimental): Oral 5-Azacitidine 100 mg (Days 1-14) Romidepsin (10 mg/m2, Days 8 and 15), cycle length (28 days)
  Interventions: Drug: RomiDEPsin 10 MG/M2; Drug: Oral 5-Azacitidine 100 MG
- R/O: Level 2 (Experimental): Oral 5-Azacitidine 200 mg (Days 1-14) Romidepsin (10 mg/m2, Days 8 and 15), cycle length (28 days)
  Interventions: Drug: RomiDEPsin 10 MG/M2; Drug: Oral 5-Azacitidine 200 MG
- R/O: Level 3 (Experimental): Oral 5-Azacitidine 300 mg (Days 1-14) Romidepsin (10 mg/m2, Days 8 and 15), cycle length (28 days)
  Interventions: Drug: RomiDEPsin 10 MG/M2; Drug: Oral 5-Azacitidine 300 MG
- R/O: Level 4 (Experimental): Oral 5-Azacitidine 300 mg (Days 1-14) Romidepsin (14 mg/m2, Days 8 and 15), cycle length (28 days)
  Interventions: Drug: Romidepsin 14 MG/M2; Drug: Oral 5-Azacitidine 300 MG
- R/O: Level 5 (Experimental): Oral 5-Azacitidine 300 mg (Days 1-14) Romidepsin (14 mg/m2, Days 8, 15 and 22), cycle length (35 days)
  Interventions: Drug: Romidepsin 14 MG/M2; Drug: Oral 5-Azacitidine 300 MG
- R/O: Level 6 (Experimental): Oral 5-Azacitidine 300 mg (Days 1-21) Romidepsin (14 mg/m2, Days 8, 15 and 22), cycle length (35 days)
  Interventions: Drug: Romidepsin 14 MG/M2; Drug: Oral 5-Azacitidine 300 MG

INTERVENTIONS:
Drug: RomiDEPsin 10 MG/M2 — Romidepsin is an anti-cancer ("antineoplastic" or "cytotoxic") chemotherapy drug. Romidepsin is classified as a "Histone Deacetylase Inhibitor".
  Dose escalation (10 mg/m2)
  Other Names: Istodax
  Arms: R/O: Level -1; R/O: Level 1; R/O: Level 2; R/O: Level 3
Drug: Oral 5-Azacitidine 100 MG — A pyrimidine nucleoside analogue of cytidine with antineoplastic activity.
  Dose escalation (100 mg)
  Other Names: 5-AC
  Arms: R/O: Level -1; R/O: Level 1
Drug: Romidepsin 14 MG/M2 — Romidepsin is an anti-cancer ("antineoplastic" or "cytotoxic") chemotherapy drug. Romidepsin is classified as a "Histone Deacetylase Inhibitor".
  Dose escalation (14 mg/m2)
  Other Names: Istodax
  Arms: R/O: Level 4; R/O: Level 5; R/O: Level 6
Drug: Oral 5-Azacitidine 200 MG — A pyrimidine nucleoside analogue of cytidine with antineoplastic activity.
  Dose escalation (200 mg)
  Other Names: 5-AC
  Arms: R/O: Level 2
Drug: Oral 5-Azacitidine 300 MG — A pyrimidine nucleoside analogue of cytidine with antineoplastic activity.
  Dose escalation (300 mg)
  Other Names: 5-AC
  Arms: R/O: Level 3; R/O: Level 4; R/O: Level 5; R/O: Level 6

SUMMARY:
This is an open label, phase I/IIa, 3 x 3 dose escalation study with an initial phase I followed by a disease focused phase II.

The primary objective of the phase I is to determine the maximum tolerated dose (MTD) and dose limiting toxicity (DLT) of the combinations of oral 5-azacitidine and romidepsin in patients with lymphoma. The safety and toxicity of this combination will be evaluated throughout the entire study.

If the combination of oral 5-azacitidine and romidepsin is found to be feasible and an MTD is established, the phase II part of the study will be initiated.

Phase II will consist of a 2 stage design of the combination of oral 5-azacitidine and romidepsin for patients with relapsed or refractory T-cell lymphomas.

DETAILED DESCRIPTION:
Subjects will receive oral 5-azacitidine and romidepsin, administered as follows: oral 5-azacitidine from Days 1-14 (Dose cohorts -1 to 5) or Days 1-21 (Dose cohort 6); and romidepsin administered intravenously on Days 8 (Dose cohorts 1-4) of a 28 day cycle, and Day 22 (Dose cohorts 5 and 6) of a 35 day cycle. Cohorts of 3 patients will be enrolled sequentially as outlined in the dose escalation scheme. Once the MTD is reached the Phase II part of the protocol will be initiated in patients with T-Cell Lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Phase I: Histologically confirmed relapsed or refractory non-Hodgkin lymphoma or Hodgkin lymphoma (WHO criteria), with no accepted curative options.
* Phase II: Relapsed or refractory T-cell lymphoma, including patients with central nervous system (CNS) involvement or lymphomatous meningitis are allowed on study.
* Relapsed or refractory disease following frontline chemotherapy. No upper limit for the number of prior therapies. Patients may have relapsed after prior autologous or allogeneic stem cell transplant.
* Evaluable Disease in the Phase I, and measurable disease for the Phase II.
* Age > or = 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status < or = 2.
* Patients must have adequate organ and marrow function.
* Negative urine or serum pregnancy test for females of childbearing potential.
* All females of childbearing potential must use an effective barrier method of contraception during the treatment period and for at least 1 month thereafter. Male subjects should use a barrier method of contraception during the treatment period and for at least 3 months thereafter.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior Therapy

  * Exposure to chemotherapy or radiotherapy within 2 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 2 weeks earlier.
  * Systemic steroids that have not been stabilized ( ≥ 5 days) to the equivalent of ≤10 mg/day prednisone prior to the start of the study drugs.
  * No other concurrent investigational agents are allowed.
* History of allergic reactions to Oral 5-azacitidine or Romidepsin.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women.
* Nursing women.
* Active concurrent malignancy (except non-melanoma skin cancer or carcinoma in situ of the cervix). If there is a history of prior malignancy, the patient must be disease-free for ≥ 3 years.
* Patients known to be Human Immunodeficiency Virus (HIV)-positive.
* Patients with active hepatitis A, hepatitis B, or hepatitis C infection.
* Concomitant use of CYP3A4 inhibitors.
* Any known cardiac abnormalities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2020-01-06 (Actual); Study Completion 2020-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Owen A. O'Connor, MD, Ph.D., Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Falchi L, Ma H, Klein S, Lue JK, Montanari F, Marchi E, Deng C, Kim HA, Rada A, Jacob AT, Kinahan C, Francescone MM, Soderquist CR, Park DC, Bhagat G, Nandakumar R, Menezes D, Scotto L, Sokol L, Shustov AR, O'Connor OA. Combined oral 5-azacytidine and romidepsin are highly effective in patients with PTCL: a multicenter phase 2 study. Blood. 2021 Apr 22;137(16):2161-2170. doi: 10.1182/blood.2020009004. PMID 33171487
- [Derived] O'Connor OA, Falchi L, Lue JK, Marchi E, Kinahan C, Sawas A, Deng C, Montanari F, Amengual JE, Kim HA, Rada AM, Khan K, Jacob AT, Malanga M, Francescone MM, Nandakumar R, Soderquist CR, Park DC, Bhagat G, Cheng B, Risueno A, Menezes D, Shustov AR, Sokol L, Scotto L. Oral 5-azacytidine and romidepsin exhibit marked activity in patients with PTCL: a multicenter phase 1 study. Blood. 2019 Oct 24;134(17):1395-1405. doi: 10.1182/blood.2019001285. PMID 31471376

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From November 2013 through January 2016, 33 patients were enrolled, and 7 withdrew from the study before receiving the study interventions. 26 patients received the study interventions in Phase 1. From April 2017 and March 2019, 25 patients were enrolled in Phase 2 and received the study interventions.
Pre-assignment Details: The participants in Phase 1 (n=26) are a different population than the participants in Phase 2 (n=25).
Groups:
- Phase 1, Dose Level 1: Oral 5-Azacitidine 100 mg and Romidepsin 10 mg/m2: Cohort 1: Participants were administered 100 mg of oral 5-Azacitidine (Days 1-14) and 10 mg/m2 of Romidepsin (Days 8 and 15) every 21 days
- Phase 1, Dose Level 2: Oral 5-Azacitidine 200 mg and Romidepsin 10 mg/m2: Cohort 2: Participants were administered 200 mg of oral 5-Azacitidine (Days 1-14) and 10 mg/m2 of Romidepsin (Days 8 and 15) every 21 days
- Phase 1, Dose Level 3: Oral 5-Azacitidine 200 mg and Romidepsin 10 mg/m2 (Extended Cycle): Cohort 3: Participants were administered 200 mg of oral 5-Azacitidine (Days 1-14) and 10 mg/m2 of Romidepsin (Days 8 and 15) every 28 days
- Phase 1, Dose Level 4: Oral 5-Azacitidine 300 mg and Romidepsin 10 mg/m2: Cohort 4: Participants were administered 300 mg of oral 5-Azacitidine (Days 1-14) and 10 mg/m2 of Romidepsin (Days 8 and 15) every 28 days
- Phase 1, Dose Level 5: Oral 5-Azacitidine 300 mg and Romidepsin 14 mg/m2: Cohort 5: Participants were administered 300 mg of oral 5-Azacitidine (Days 1-14) and 14 mg/m2 of Romidepsin (Days 8, 15, and 22) every 28 days
- Phase 1, Dose Level 6: Oral 5-Azacitidine 300 mg and Romidepsin 14 mg/m2: Cohort 6: Participants were administered 300 mg of oral 5-Azacitidine (Days 1-14) and 14mg/m2 of Romidepsin (Days 8, 15, and 22) every 35 days.
  Determined to be the Maximum Tolerated Dose (MTD) i.e. the Recommended Phase 2 Dose (RP2D)
- Phase 1, Dose Level 6 (MTD): Oral 5-Azacitidine 300 mg and Romidepsin 14 mg/m2: Expanded Cohort 6: Participants were administered 300 mg of oral 5-Azacitidine (Days 1-21) and 14 mg/m2 of Romidepsin (Days 8, 15, and 22) every 35 days.
  Determined to be the MTD (Maximum Administrable Dose)
- Phase 2, MTD: Oral 5-Azacitidine 300 mg and Romidepsin 14 mg/m2: Patients will be treated with oral 5-azacytidine and Romidepsin at the MTD. The treatment will be administered as follows: oral 5-azacytidine 300 mg (flat dose) on Days 1-14 and Romidepsin 14 mg/m2 (flat dose) on Days 8, 15, and 22 on a 35-day cycle.
Period: Phase 1: Dose Level 1
Arm/Group | Phase 1, Dose Level 1: Oral 5-Azacitidine 100 mg and Romidepsin 10 mg/m2 | Phase 1, Dose Level 2: Oral 5-Azacitidine 200 mg and Romidepsin 10 mg/m2 | Phase 1, Dose Level 3: Oral 5-Azacitidine 200 mg and Romidepsin 10 mg/m2 (Extended Cycle) | Phase 1, Dose Level 4: Oral 5-Azacitidine 300 mg and Romidepsin 10 mg/m2 | Phase 1, Dose Level 5: Oral 5-Azacitidine 300 mg and Romidepsin 14 mg/m2 | Phase 1, Dose Level 6: Oral 5-Azacitidine 300 mg and Romidepsin 14 mg/m2 | Phase 1, Dose Level 6 (MTD): Oral 5-Azacitidine 300 mg and Romidepsin 14 mg/m2 | Phase 2, MTD: Oral 5-Azacitidine 300 mg and Romidepsin 14 mg/m2
Started | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 1: Dose Level 2
Arm/Group | Phase 1, Dose Level 1: Oral 5-Azacitidine 100 mg and Romidepsin 10 mg/m2 | Phase 1, Dose Level 2: Oral 5-Azacitidine 200 mg and Romidepsin 10 mg/m2 | Phase 1, Dose Level 3: Oral 5-Azacitidine 200 mg and Romidepsin 10 mg/m2 (Extended Cycle) | Phase 1, Dose Level 4: Oral 5-Azacitidine 300 mg and Romidepsin 10 mg/m2 | Phase 1, Dose Level 5: Oral 5-Azacitidine 300 mg and Romidepsin 14 mg/m2 | Phase 1, Dose Level 6: Oral 5-Azacitidine 300 mg and Romidepsin 14 mg/m2 | Phase 1, Dose Level 6 (MTD): Oral 5-Azacitidine 300 mg and Romidepsin 14 mg/m2 | Phase 2, MTD: Oral 5-Azacitidine 300 mg and Romidepsin 14 mg/m2
Started | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 1: Dose Level 3
Arm/Group | Phase 1, Dose Level 1: Oral 5-Azacitidine 100 mg and Romidepsin 10 mg/m2 | Phase 1, Dose Level 2: Oral 5-Azacitidine 200 mg and Romidepsin 10 mg/m2 | Phase 1, Dose Level 3: Oral 5-Azacitidine 200 mg and Romidepsin 10 mg/m2 (Extended Cycle) | Phase 1, Dose Level 4: Oral 5-Azacitidine 300 mg and Romidepsin 10 mg/m2 | Phase 1, Dose Level 5: Oral 5-Azacitidine 300 mg and Romidepsin 14 mg/m2 | Phase 1, Dose Level 6: Oral 5-Azacitidine 300 mg and Romidepsin 14 mg/m2 | Phase 1, Dose Level 6 (MTD): Oral 5-Azacitidine 300 mg and Romidepsin 14 mg/m2 | Phase 2, MTD: Oral 5-Azacitidine 300 mg and Romidepsin 14 mg/m2
Started | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 1: Dose Level 4
Arm/Group | Phase 1, Dose Level 1: Oral 5-Azacitidine 100 mg and Romidepsin 10 mg/m2 | Phase 1, Dose Level 2: Oral 5-Azacitidine 200 mg and Romidepsin 10 mg/m2 | Phase 1, Dose Level 3: Oral 5-Azacitidine 200 mg and Romidepsin 10 mg/m2 (Extended Cycle) | Phase 1, Dose Level 4: Oral 5-Azacitidine 300 mg and Romidepsin 10 mg/m2 | Phase 1, Dose Level 5: Oral 5-Azacitidine 300 mg and Romidepsin 14 mg/m2 | Phase 1, Dose Level 6: Oral 5-Azacitidine 300 mg and Romidepsin 14 mg/m2 | Phase 1, Dose Level 6 (MTD): Oral 5-Azacitidine 300 mg and Romidepsin 14 mg/m2 | Phase 2, MTD: Oral 5-Azacitidine 300 mg and Romidepsin 14 mg/m2
Started | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 1: Dose Level 5
Arm/Group | Phase 1, Dose Level 1: Oral 5-Azacitidine 100 mg and Romidepsin 10 mg/m2 | Phase 1, Dose Level 2: Oral 5-Azacitidine 200 mg and Romidepsin 10 mg/m2 | Phase 1, Dose Level 3: Oral 5-Azacitidine 200 mg and Romidepsin 10 mg/m2 (Extended Cycle) | Phase 1, Dose Level 4: Oral 5-Azacitidine 300 mg and Romidepsin 10 mg/m2 | Phase 1, Dose Level 5: Oral 5-Azacitidine 300 mg and Romidepsin 14 mg/m2 | Phase 1, Dose Level 6: Oral 5-Azacitidine 300 mg and Romidepsin 14 mg/m2 | Phase 1, Dose Level 6 (MTD): Oral 5-Azacitidine 300 mg and Romidepsin 14 mg/m2 | Phase 2, MTD: Oral 5-Azacitidine 300 mg and Romidepsin 14 mg/m2
Started | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 1: Dose Level 6
Arm/Group | Phase 1, Dose Level 1: Oral 5-Azacitidine 100 mg and Romidepsin 10 mg/m2 | Phase 1, Dose Level 2: Oral 5-Azacitidine 200 mg and Romidepsin 10 mg/m2 | Phase 1, Dose Level 3: Oral 5-Azacitidine 200 mg and Romidepsin 10 mg/m2 (Extended Cycle) | Phase 1, Dose Level 4: Oral 5-Azacitidine 300 mg and Romidepsin 10 mg/m2 | Phase 1, Dose Level 5: Oral 5-Azacitidine 300 mg and Romidepsin 14 mg/m2 | Phase 1, Dose Level 6: Oral 5-Azacitidine 300 mg and Romidepsin 14 mg/m2 | Phase 1, Dose Level 6 (MTD): Oral 5-Azacitidine 300 mg and Romidepsin 14 mg/m2 | Phase 2, MTD: Oral 5-Azacitidine 300 mg and Romidepsin 14 mg/m2
Started | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 1: Dose Level 6 (Expanded Cohort)
Arm/Group | Phase 1, Dose Level 1: Oral 5-Azacitidine 100 mg and Romidepsin 10 mg/m2 | Phase 1, Dose Level 2: Oral 5-Azacitidine 200 mg and Romidepsin 10 mg/m2 | Phase 1, Dose Level 3: Oral 5-Azacitidine 200 mg and Romidepsin 10 mg/m2 (Extended Cycle) | Phase 1, Dose Level 4: Oral 5-Azacitidine 300 mg and Romidepsin 10 mg/m2 | Phase 1, Dose Level 5: Oral 5-Azacitidine 300 mg and Romidepsin 14 mg/m2 | Phase 1, Dose Level 6: Oral 5-Azacitidine 300 mg and Romidepsin 14 mg/m2 | Phase 1, Dose Level 6 (MTD): Oral 5-Azacitidine 300 mg and Romidepsin 14 mg/m2 | Phase 2, MTD: Oral 5-Azacitidine 300 mg and Romidepsin 14 mg/m2
Started | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 2: MTD
Arm/Group | Phase 1, Dose Level 1: Oral 5-Azacitidine 100 mg and Romidepsin 10 mg/m2 | Phase 1, Dose Level 2: Oral 5-Azacitidine 200 mg and Romidepsin 10 mg/m2 | Phase 1, Dose Level 3: Oral 5-Azacitidine 200 mg and Romidepsin 10 mg/m2 (Extended Cycle) | Phase 1, Dose Level 4: Oral 5-Azacitidine 300 mg and Romidepsin 10 mg/m2 | Phase 1, Dose Level 5: Oral 5-Azacitidine 300 mg and Romidepsin 14 mg/m2 | Phase 1, Dose Level 6: Oral 5-Azacitidine 300 mg and Romidepsin 14 mg/m2 | Phase 1, Dose Level 6 (MTD): Oral 5-Azacitidine 300 mg and Romidepsin 14 mg/m2 | Phase 2, MTD: Oral 5-Azacitidine 300 mg and Romidepsin 14 mg/m2
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 25
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 25
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics and study results were only collected as the combined total from participants per study phase. Baseline characteristics were not collected per dose level and thus cannot be reported per dose level.
  Baseline characteristics were collected from all participants who enrolled/consented in Phase 1 (n=33) and Phase 2 (n=25). Of those 33 enrolled in Phase 1, 26 received the study interventions and only those 26 are counted in the Participant Flow.
Groups:
- Phase 1: Phase 1 is to determine the maximum tolerated dose (MTD) and dose limiting toxicity (DLT) of the combinations of oral 5-azacitidine and romidepsin in patients with lymphoma. Patients will be administered the study drugs in a 3 + 3 dose-escalation study.
- Phase 2: Patients will be treated with oral 5-azacytidine and Romidepsin at the MTD. The treatment will be administered as follows: oral 5-azacytidine 300 mg (flat dose) on Days 1-14 and Romidepsin 14 mg/m2 (flat dose) on Days 8, 15, and 22 on a 35-day cycle.
- Total: Total of all reporting groups
Arm/Group | Phase 1 | Phase 2 | Total
Number analyzed (Participants) | 33 | 25 | 58
Age, Continuous [Median (Full Range); unit: years] | 57 [23 to 79] | 63 [42 to 88] | NA [23 to 88] — The median age for the entire study was not calculated at the time of data analysis. The standard deviation cannot be calculated without the raw data. The raw data cannot be accessed, as the Principal Investigator and entire study team has left the institution. In addition, the study closed with the Institutional Review Board in 2021 and further analysis cannot be conducted.
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 19 | 15 | 34
  Unknown | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 3 | 13
  Not Hispanic or Latino | 20 | 22 | 42
  Unknown or Not Reported | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 1 | 6
  White | 25 | 22 | 47
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Maximum Tolerated Dose (MTD) of the Combination of Oral 5-azacitidine in Combination With Romidepsin
Description: The highest dose of a drug or treatment that does not cause unacceptable side effects. The MTD is determined in clinical trials by testing increasing doses on different groups of people until the highest dose with acceptable side effects is found.
Time Frame: up to 1.5 years
Population: This Outcome Measure is specific for Phase 1 of the study. This Outcome Measure was NOT applied to Phase 2, therefore data was only collected and reported for Phase 1.
  26 participants received the study interventions in Phase 1.
Measure: Number; unit: mg
Groups:
- Phase I: Phase I is to determine the maximum tolerated dose (MTD) and dose limiting toxicity (DLT) of the combinations of oral 5-azacitidine and romidepsin in patients with lymphoma. The safety and toxicity of this combination will be evaluated throughout the entire study.
Arm/Group | Phase I
Number analyzed (Participants) | 26
mg | 300

2. Primary Outcome: Phase I: Maximum Tolerated Dose (MTD) of Romidepsin in Combination With Oral 5-azacytidine
Description: as for outcome 1
Time Frame: up to 1.5 years
Population: as for outcome 1
Measure: Number; unit: mg/m2
Arm/Group | Phase I
Number analyzed (Participants) | 26
mg/m2 | 14

3. Primary Outcome: Percentage of Patients Who Experienced Significant Toxicities in Phase 1
Description: Patients receiving the combination of oral 5-azacitidine and romidepsin and experiencing grades 1-4 toxicities will be tallied based on events observed and assessed by a qualified investigator. This Outcome Measure is specifically for Phase 1 of the study.
Time Frame: Up to 1.5 years
Population: This Outcome Measure is specific for Phase 1 of the study. This Outcome Measure was NOT applied to Phase 2, therefore data was only collected and reported for Phase 1. Results were not collected per dose level and thus cannot be reported per dose level.
  26 participants received the study interventions in Phase 1.
Measure: Number; unit: percentage of participants
Arm/Group | Phase I
Number analyzed (Participants) | 26
percentage of participants | 10

4. Primary Outcome: Phase II: Overall Response Rate (ORR) (Complete + Partial Response) of the Combination of Oral 5-azacitidine and Romidepsin in Patients With Relapsed/Refractory T-Cell Lymphoma
Description: The percentage of people in a study or treatment group who have a partial response or complete response to the treatment within a certain period of time. A partial response is a decrease in the size of a tumor or in the amount of cancer in the body, and a complete response is the disappearance of all signs of cancer in the body. In a clinical trial, measuring the ORR is one way to see how well a new treatment works.
Time Frame: Up to 3 years
Population: This Outcome Measure is specific for Phase 2 of the study, therefore data was only collected and reported for Phase 2. Results were not collected per dose level and thus cannot be reported per dose level.
Measure: Number; unit: percentage of participants
Groups:
- Phase II: Patients will be treated with oral 5-azacytidine and romidepsin at the MTD. The treatment will be administered as follows: oral 5azacytidine 300 mg (flat dose) Days 1-14 and romidepsin 14 mg/m2 on Days 8, 15, and 22 on an every 35 day cycle.
Arm/Group | Phase II
Number analyzed (Participants) | 25
percentage of participants | 30

ADVERSE EVENTS:
Time Frame: 1.5 years
Description: Adverse events were only recorded/collected as the combined total from participants per study phase. Adverse events were not collected per dose level and thus cannot be reported per dose level.
  For Phase 1, adverse events were collected from the 26 participants who received the study interventions and completed the study.
Groups:
- Phase 1: Phase 1 is to determine the maximum tolerated dose (MTD) and dose limiting toxicity (DLT) of the combinations of oral 5-azacitidine and romidepsin in patients with lymphoma. Patients will be administered the study drugs in a 3 + 3 dose-escalation study.
  Romidepsin is an anti-cancer ("antineoplastic" or "cytotoxic") chemotherapy drug. Romidepsin is classified as a "Histone Deacetylase Inhibitor". Dose escalation: 10, 14 mg/m2
  Oral 5-Azacitidine is a pyrimidine nucleoside analogue of cytidine with antineoplastic activity. Dose escalation: 100, 200, 300 mg
Arm/Group | Phase 1 | Phase 2
All-Cause Mortality (participants affected / at risk) | 11/26 | 0/25
Serious Adverse Events (participants affected / at risk) | 11/26 | 12/25
Other Adverse Events (participants affected / at risk) | 26/26 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 (N=26) | Phase 2 (N=25)
Alkaline phosphatase elevation (General disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 5 | 4
Febrile neutropenia (General disorders) | 2 | 3
Hyperglycemia (Grade 3 and 4) (Endocrine disorders) | 1 | 1
Hypermagnesemia (Renal and urinary disorders) | 1 | 0
Hypokalemia (General disorders) | 1 | 0
Hyponatremia (General disorders) | 2 | 0
Hypotension (General disorders) | 3 | 0
Lymphocyte count decrease (Immune system disorders) | 11 | 8
Neutrophil count decrease (Immune system disorders) | 11 | 10
Platelet count decrease (Immune system disorders) | 7 | 12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 (N=26) | Phase 2 (N=25)
Fatigue (General disorders) | 10 | 13
Nausea (General disorders) | 14 | 15
Vomiting (General disorders) | 12 | 10
Creatinine elevation (Renal and urinary disorders) | 8 | 10
Diarrhea (Gastrointestinal disorders) | 7 | 12
Fever (General disorders) | 3 | 7
Hypercalcemia (Blood and lymphatic system disorders) | 3 | 3
Hypoalbuminemia (General disorders) | 13 | 11
Hypocalcemia (Blood and lymphatic system disorders) | 5 | 7
Hypoglycemia (General disorders) | 3 | 3
Hyperglycemia (Grade 1 and 2) (Endocrine disorders) | 21 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-20): https://cdn.clinicaltrials.gov/large-docs/35/NCT01998035/Prot_SAP_000.pdf